CLINICAL TRIAL: NCT04053842
Title: Multi-modality Prostate Cancer Image Guided Interventions - 5
Brief Title: Multi-modality Imaging (PCa) Using Sodium MRI and PSMA PET in Men Pre-prostatectomy
Acronym: IGPC-5
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Glenn Bauman (Other)
Collaborators: Western University, Canada (Other); United States Department of Defense (U.S. Federal Agency); Centre for Probe Development and Commercialization (Other)
Responsible Party: Sponsor-Investigator, Glenn Bauman, Overall Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Organization: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IGPC-5; REB File # 114138 (Other: Western University, Health Sciences Research Ethics Board)
Record Dates: First submitted 2019-08-08; First posted 2019-08-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Prostate Cancer; Prostate Adenocarcinoma; Prostate Neoplasm
Keywords: Prostate Cancer; PSMA PET; [18F]PSMA-1007 PET/CT imaging; Radical Prostatectomy; Sodium MRI; Sodium Imaging
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Positron-Emission Tomography; Multiparametric Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Multi-modality prostate cancer imaging (Experimental): The study requires eligible patients to complete one imaging session at St. Joseph's Health Care to begin within 6 weeks of the scheduled Radical Prostatectomy. Imaging will consist of simultaneous multiparametric MRI (mpMRI), sodium MRI and positron emission tomography (PET) with a radio-labeled probe for prostate-specific membrane antigen (PSMA).
  Interventions: Diagnostic Test: PET Scan; Drug: [18F]PSMA-1007 Injection; Diagnostic Test: Sodium MRI; Diagnostic Test: Multiparametric MRI

INTERVENTIONS:
Diagnostic Test: PET Scan — PET imaging uses small amounts of a radioactive substance called a tracer to look for disease in the body. The radioactive substance used in this study is [18F]PSMA-1007.
  Other Names: PSMA PET
Drug: [18F]PSMA-1007 Injection — [18F]PSMA-1007 is given by intravenous (IV) injection into the arm. It travels through the blood stream where it is rapidly taken up by prostate cancer cells and emits tiny, positively charged particles (called positrons) that produce signals into the body. These signals are detected by the PET component of the PET/MRI scanner.
  Other Names: PSMA
Diagnostic Test: Sodium MRI — Sodium MRI uses magnetic waves and a specially-designed rectal probe to measure the sodium concentration (amount of salt) in the prostate. Previous research has shown that higher sodium concentrations in the prostate might be a sign of more aggressive cancer.
Diagnostic Test: Multiparametric MRI — MRI is a common medical diagnostic tool that uses magnetic waves and a contrast agent (dye) called Gadovist to take pictures of body tissue.
  Other Names: mpMRI

SUMMARY:
The study is a non-randomized, prospective trial of men scheduled for radical prostatectomy for treatment of prostate cancer as standard of care and will undergo a series of pre-operative multi-modality imaging studies. Pre-operative imaging will be correlated with actual pathology results and statistical modeling performed to determine the most informative imaging biomarkers in predicting cancer location and aggressiveness (Gleason Score).

DETAILED DESCRIPTION:
The over-arching goal is to "improve the quality of life for survivors of prostate cancer" through advanced imaging tools for improved pre-treatment detection and characterization of prostate cancer through non-invasive imaging.

Seminal research measuring tissue sodium concentration (TSC) in human PCa with sodium MRI has demonstrated increased TSC in prostate lesions related to tumor aggressiveness. This suggests that the addition of sodium MRI to mpMRI data will enhance the identification and characterization of prostate lesions in men with PCa. This will improve the healthcare of men through better risk stratification and treatment decisions, which will ultimately reduce overtreatment. Radio-labeled PET tracers that target PSMA have demonstrated exceptional sensitivity for molecular imaging of prostate lesions. Lesion-detection specificity of combined PSMA PET and mpMRI is very high (97 - 100%). However, PSMA PET is not practical for active surveillance of prostate cancer within the current healthcare system due to limited access and the fact that its added cost and radiation dose restricts its utility for repeated scans. However, as a tool to develop and validate our imaging assay, it is unparalleled. Compared with hybrid PET/MRI, a single modality imaging assay based only on mpMRI contrasts and endogenous TSC would be more widely available, cost effective and find wider clinical adoption - particularly for AS. The immediate expected outcome from this project is that an MRI assay combining data from mpMRI and sodium MRI will have a similar ability as PSMA PET to accurately discriminate between low- and high-risk PCa for improved treatment decisions and surveillance of low-risk disease.

The transformative potential of a non-invasive, single modality, whole-gland imaging assay comprised of biomarkers from combined TSC and mpMRI could ultimately replace serial biopsies for surveillance of men with low- and intermediate-risk disease. Patients who are educated to understand the typical slow progression of low-risk PCa, surveillance methods and treatment risks are more likely to consider AS. In a systematic approach developed to improve physician counselling of low-risk PCa patients, the acceptance rate for AS was improved to 94% - a relative reduction of approximately 30% in the risk of unnecessary curative treatment. However, it is also important to note that the rate of subsequent treatment for men undergoing AS may be as high as 50% over 10 years of follow-up. The majority of these men are transitioned to treatment within 2-3 years of initial diagnosis. Identification of those men who fit the criteria for AS but are destined to have early progression is an important clinical goal. Those men can be streamed to early treatment through longitudinal assessment of lesion progression with this imaging assay and thus increase the confidence and uptake of AS protocols. AS of PCa (including possible delayed treatment) saves costs over the lifetime of a patient, compared with immediate treatment and provides superior quality of life.

Research Strategy: The investigators will evaluate a non-invasive imaging assay for in vivo characterization of prostate lesions comprised of clinical multi-parametric magnetic resonance imaging (mpMRI) combined with sodium magnetic resonance imaging (sodium MRI) in a cohort of men with biopsy-proven prostate cancer. The use of mpMRI to detect, localize and stage prostate cancer is becoming standard clinical practice. Prior research in ten patients has established that tissue sodium concentration (TSC) assessed by sodium MRI increases significantly with histological grade in prostate lesions. The addition of TSC data to conventional mpMRI data (i.e. ADC values, T2 contrast, contrast agent wash-in/out rates) will be evaluated in a multivariate data analysis to demonstrate that a combination of these imaging protocols improves the characterization of PCa. The resulting predictive tool (imaging assay) will accurately discriminate between low- and high-risk PCa for improved treatment decisions and to assess possible progression of low-risk disease during surveillance.

This imaging assay will be validated against positron emission tomography (PET) using a radio-labeled tracer which binds to prostate-specific membrane antigen (PSMA). PSMA PET is arguably the most sensitive imaging method for detection of intra-prostatic lesions. Importantly, it has a high sensitivity for prostate lesion detection (>90%), even for lower tumor grades where mpMRI has difficulties. Maximum standard uptake value (SUVmax) of this radiotracer has been positively correlated with Gleason grade and as such, is an excellent comparator for TSC assessment of lesion aggressiveness. Unfortunately, the limited accessibility and cost of PET hinders its clinical application.

In this project, the investigators expect to validate that the addition of sodium MRI to mpMRI can provide similar lesion characterization compared to PSMA PET. Data supporting this hypothesis will be acquired using a hybrid PET/MRI system because this is the best imaging platform for this project. If successful, the incorporation of sodium MRI into existing mpMRI protocols would improve characterization of disease and be a more cost effective and generalizable innovation compared to PET-based techniques that require both an expensive probe as well as hybrid imaging platforms.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent for this study
* Male, aged 18 years or older
* Pathologically confirmed prostate cancer on previous biopsy
* Suitable for and consenting to Radical Prostatectomy for treatment as standard of care

Exclusion Criteria:

* Prior therapy for prostate cancer (including hormone therapy)
* Use of 5-alpha reductase inhibitors, i.e. finasteride (Proscar) or dutasteride (Avodart) within 6 months of study start. Patients undergoing a 6-month washout period prior to study start will be eligible.
* Inability to comply with the pre-operative imaging panel
* Patients scheduled for radical prostatectomy with prostate size exceeding 65 cc
* Allergy to contrast agents to be used as part of the imaging panel
* Acute kidney injury (AKI), chronic kidney disease (CKD) Stage 4 or 5 (estimated Glomerular Filtration Rate [eGFR] < 30 mL/min/1.73m2) or those on dialysis
* Post-void residual urine volume > 150 cc (determined by post-void ultrasound)
* Hip prosthesis, vascular grafting that is MRI incompatible or sources of artefact within the pelvis
* Contraindication to MRI

  * pacemaker or other electronic implants
  * known metal in the orbit
  * cerebral aneurysm clips

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate cancer is a male disease.
Enrollment: 45 (Estimated)
Dates: Start 2021-02-04 (Actual); Primary Completion 2024-01-23 (Actual); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Pathologic Validation and Modeling | 4 years
  We will evaluate the ability of simultaneous multiparametric MRI (mpMRI), sodium MRI and positron emission tomography (PET) with a radio-labeled probe for prostate-specific membrane antigen (PSMA) to accurately predict the actual cancer distribution found in the whole mount prostatectomy specimens obtained from the surgery.
  A variety of statistical methods will be utilized to build predictive models based on the extracted features and to identify a final model that will be used as the predictive tool (i.e. the imaging assay).
  We will quantify the ability of these models to enhance clinical lesion identification.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Pautler, MD, FRCSC, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chun FK, Karakiewicz PI, Briganti A, Walz J, Kattan MW, Huland H, Graefen M. A critical appraisal of logistic regression-based nomograms, artificial neural networks, classification and regression-tree models, look-up tables and risk-group stratification models for prostate cancer. BJU Int. 2007 Apr;99(4):794-800. doi: 10.1111/j.1464-410X.2006.06694.x. PMID 17378842
- [Background] Makarov DV, Trock BJ, Humphreys EB, Mangold LA, Walsh PC, Epstein JI, Partin AW. Updated nomogram to predict pathologic stage of prostate cancer given prostate-specific antigen level, clinical stage, and biopsy Gleason score (Partin tables) based on cases from 2000 to 2005. Urology. 2007 Jun;69(6):1095-101. doi: 10.1016/j.urology.2007.03.042. PMID 17572194
- [Background] Hricak H, Choyke PL, Eberhardt SC, Leibel SA, Scardino PT. Imaging prostate cancer: a multidisciplinary perspective. Radiology. 2007 Apr;243(1):28-53. doi: 10.1148/radiol.2431030580. PMID 17392247
- [Background] Chan I, Wells W 3rd, Mulkern RV, Haker S, Zhang J, Zou KH, Maier SE, Tempany CM. Detection of prostate cancer by integration of line-scan diffusion, T2-mapping and T2-weighted magnetic resonance imaging; a multichannel statistical classifier. Med Phys. 2003 Sep;30(9):2390-8. doi: 10.1118/1.1593633. PMID 14528961
- [Background] Barrett T, Turkbey B, Choyke PL. PI-RADS version 2: what you need to know. Clin Radiol. 2015 Nov;70(11):1165-76. doi: 10.1016/j.crad.2015.06.093. Epub 2015 Jul 29. PMID 26231470
- [Background] Kwee SA, Thibault GP, Stack RS, Coel MN, Furusato B, Sesterhenn IA. Use of step-section histopathology to evaluate 18F-fluorocholine PET sextant localization of prostate cancer. Mol Imaging. 2008 Jan-Feb;7(1):12-20. PMID 18384719
- [Background] Ward AD, Crukley C, McKenzie CA, Montreuil J, Gibson E, Romagnoli C, Gomez JA, Moussa M, Chin J, Bauman G, Fenster A. Prostate: registration of digital histopathologic images to in vivo MR images acquired by using endorectal receive coil. Radiology. 2012 Jun;263(3):856-64. doi: 10.1148/radiol.12102294. Epub 2012 Apr 2. PMID 22474671
- [Background] Han W, Johnson C, Gaed M, Gomez JA, Moussa M, Chin JL, et al. Automatic cancer detection and localization on prostatectomy histopathology images. In: Tomaszewski JE, Gurcan MN, editors. Medical Imaging 2018: Digital Pathology. Proceedings of SPIE. 10581. Bellingham: Spie-Int Soc Optical Engineering; 2018
- [Background] Alfano R, Soetemans D, Bauman GS, Gibson E, Gaed M, Moussa M, et al. Development of a Computer Aided Diagnosis Model for Prostate Cancer Classification on Multi-Parametric MRI. In: Petrick N, Mori K, editors. Medical Imaging 2018: Computer-Aided Diagnosis. Proceedings of SPIE. 10575. Bellingham: Spie-Int Soc Optical Engineering; 2018.
- [Background] Evans JD, Jethwa KR, Ost P, Williams S, Kwon ED, Lowe VJ, Davis BJ. Prostate cancer-specific PET radiotracers: A review on the clinical utility in recurrent disease. Pract Radiat Oncol. 2018 Jan-Feb;8(1):28-39. doi: 10.1016/j.prro.2017.07.011. Epub 2017 Jul 20. PMID 29037965
- [Background] Broeke NC, Peterson J, Lee J, Martin PR, Farag A, Gomez JA, Moussa M, Gaed M, Chin J, Pautler SE, Ward A, Bauman G, Bartha R, Scholl TJ. Characterization of clinical human prostate cancer lesions using 3.0-T sodium MRI registered to Gleason-graded whole-mount histopathology. J Magn Reson Imaging. 2019 May;49(5):1409-1419. doi: 10.1002/jmri.26336. Epub 2018 Nov 14. PMID 30430700
- [Background] Bauman G, Martin P, Thiessen JD, Taylor R, Moussa M, Gaed M, Rachinsky I, Kassam Z, Chin J, Pautler S, Lee TY, Valliant JF, Ward A. [18F]-DCFPyL Positron Emission Tomography/Magnetic Resonance Imaging for Localization of Dominant Intraprostatic Foci: First Experience. Eur Urol Focus. 2018 Sep;4(5):702-706. doi: 10.1016/j.euf.2016.10.002. Epub 2016 Oct 26. PMID 28753797
- [Background] Uprimny C, Kroiss AS, Decristoforo C, Fritz J, von Guggenberg E, Kendler D, Scarpa L, di Santo G, Roig LG, Maffey-Steffan J, Horninger W, Virgolini IJ. 68Ga-PSMA-11 PET/CT in primary staging of prostate cancer: PSA and Gleason score predict the intensity of tracer accumulation in the primary tumour. Eur J Nucl Med Mol Imaging. 2017 Jun;44(6):941-949. doi: 10.1007/s00259-017-3631-6. Epub 2017 Jan 31. PMID 28138747
- [Background] Barrett T, Riemer F, McLean MA, Kaggie J, Robb F, Tropp JS, Warren A, Bratt O, Shah N, Gnanapragasam VJ, Gilbert FJ, Graves MJ, Gallagher FA. Quantification of Total and Intracellular Sodium Concentration in Primary Prostate Cancer and Adjacent Normal Prostate Tissue With Magnetic Resonance Imaging. Invest Radiol. 2018 Aug;53(8):450-456. doi: 10.1097/RLI.0000000000000470. PMID 29969108
- [Background] Kozlowski P, Chang SD, Meng R, Madler B, Bell R, Jones EC, Goldenberg SL. Combined prostate diffusion tensor imaging and dynamic contrast enhanced MRI at 3T--quantitative correlation with biopsy. Magn Reson Imaging. 2010 Jun;28(5):621-8. doi: 10.1016/j.mri.2010.03.011. Epub 2010 Apr 13. PMID 20392586
- [Background] Ghai S, Haider MA. Multiparametric-MRI in diagnosis of prostate cancer. Indian J Urol. 2015 Jul-Sep;31(3):194-201. doi: 10.4103/0970-1591.159606. PMID 26166962
- [Background] Barentsz JO, Richenberg J, Clements R, Choyke P, Verma S, Villeirs G, Rouviere O, Logager V, Futterer JJ; European Society of Urogenital Radiology. ESUR prostate MR guidelines 2012. Eur Radiol. 2012 Apr;22(4):746-57. doi: 10.1007/s00330-011-2377-y. Epub 2012 Feb 10. PMID 22322308
- [Background] Moore CM, Giganti F, Albertsen P, Allen C, Bangma C, Briganti A, Carroll P, Haider M, Kasivisvanathan V, Kirkham A, Klotz L, Ouzzane A, Padhani AR, Panebianco V, Pinto P, Puech P, Rannikko A, Renard-Penna R, Touijer K, Turkbey B, van Poppel H, Valdagni R, Walz J, Schoots I. Reporting Magnetic Resonance Imaging in Men on Active Surveillance for Prostate Cancer: The PRECISE Recommendations-A Report of a European School of Oncology Task Force. Eur Urol. 2017 Apr;71(4):648-655. doi: 10.1016/j.eururo.2016.06.011. Epub 2016 Jun 24. PMID 27349615
- [Background] Ehdaie B, Assel M, Benfante N, Malhotra D, Vickers A. A Systematic Approach to Discussing Active Surveillance with Patients with Low-risk Prostate Cancer. Eur Urol. 2017 Jun;71(6):866-871. doi: 10.1016/j.eururo.2016.12.026. Epub 2017 Jan 24. PMID 28129893
- [Background] Hamdy FC, Donovan JL, Lane JA, Mason M, Metcalfe C, Holding P, Davis M, Peters TJ, Turner EL, Martin RM, Oxley J, Robinson M, Staffurth J, Walsh E, Bollina P, Catto J, Doble A, Doherty A, Gillatt D, Kockelbergh R, Kynaston H, Paul A, Powell P, Prescott S, Rosario DJ, Rowe E, Neal DE; ProtecT Study Group. 10-Year Outcomes after Monitoring, Surgery, or Radiotherapy for Localized Prostate Cancer. N Engl J Med. 2016 Oct 13;375(15):1415-1424. doi: 10.1056/NEJMoa1606220. Epub 2016 Sep 14. PMID 27626136
- [Background] Klotz L. Active surveillance: the Canadian experience. Curr Opin Urol. 2012 May;22(3):222-30. doi: 10.1097/MOU.0b013e328352598c. PMID 22453335
- [Background] Wibmer AG, Burger IA, Sala E, Hricak H, Weber WA, Vargas HA. Molecular Imaging of Prostate Cancer. Radiographics. 2016 Jan-Feb;36(1):142-59. doi: 10.1148/rg.2016150059. Epub 2015 Nov 20. PMID 26587888
- [Background] Sanyal C, Aprikian AG, Cury FL, Chevalier S, Dragomir A. Management of localized and advanced prostate cancer in Canada: A lifetime cost and quality-adjusted life-year analysis. Cancer. 2016 Apr 1;122(7):1085-96. doi: 10.1002/cncr.29892. Epub 2016 Feb 1. PMID 26828716
- [Background] Hoeks CM, Barentsz JO, Hambrock T, Yakar D, Somford DM, Heijmink SW, Scheenen TW, Vos PC, Huisman H, van Oort IM, Witjes JA, Heerschap A, Futterer JJ. Prostate cancer: multiparametric MR imaging for detection, localization, and staging. Radiology. 2011 Oct;261(1):46-66. doi: 10.1148/radiol.11091822. PMID 21931141
- [Background] Udovicich C, Perera M, Hofman MS, Siva S, Del Rio A, Murphy DG, Lawrentschuk N. 68Ga-prostate-specific membrane antigen-positron emission tomography/computed tomography in advanced prostate cancer: Current state and future trends. Prostate Int. 2017 Dec;5(4):125-129. doi: 10.1016/j.prnil.2017.02.003. Epub 2017 Feb 24. PMID 29188197
- [Background] Ward A, Crukley C, McKenzie C, Montreuil J, Gibson E, Gomez JA, et al. Registration of in vivo prostate magnetic resonance images to digital histopathology images. MICCAI'10 Proceedings of the 2010 international conference on Prostate cancer imaging: computer-aided diagnosis, prognosis, and intervention; Bejing, China. Berlin: Springer-Verlag; 2010
- [Background] Hambrock T, Somford DM, Huisman HJ, van Oort IM, Witjes JA, Hulsbergen-van de Kaa CA, Scheenen T, Barentsz JO. Relationship between apparent diffusion coefficients at 3.0-T MR imaging and Gleason grade in peripheral zone prostate cancer. Radiology. 2011 May;259(2):453-61. doi: 10.1148/radiol.11091409. PMID 21502392
- [Background] Hsieh FY, Bloch DA, Larsen MD. A simple method of sample size calculation for linear and logistic regression. Stat Med. 1998 Jul 30;17(14):1623-34. doi: 10.1002/(sici)1097-0258(19980730)17:143.0.co;2-s. PMID 9699234